CLINICAL TRIAL: NCT07285187
Title: Intraoperative Venous Congestion And Delirium After Cardiac Surgery: A Prospective Cohort Study
Brief Title: Venous Congestion And Delirium After Cardiac Surgery
Status: Recruiting | Type: Observational
Sponsor: Zhuan Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhuan Zhang, MD, the Deputy Director of Anesthesiology, the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou University
Organization: Yangzhou University (Other)
Other Study IDs: 20240915
Record Dates: First submitted 2024-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Intraoperative; Venous Congestion; Postoperative Delirium (POD); Cardiac Surgery
MeSH Terms: conditions — Hyperemia; Emergence Delirium | interventions — Comorbidity; Laboratories

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients scheduled to undergo elective cardiac surgery
  Interventions: Other: collection of demographic characteristics and comorbidities; Other: surgery-related parameters; Other: POD assessments; Other: collection of biological (laboratory) parameters; Other: collection of hemodynamic parameters; Other: collection of echocardiographic parameters and venous ultrasound assessments; Other: collection of parameters monitoring on the central nervous system

INTERVENTIONS:
Other: collection of demographic characteristics and comorbidities — 1. gender, age, BMI, ASA classification, NYHA (New York Heart Association) classification, MMSE score.
  2. smoking history, medical history (hypertension, diabetes mellitus, Hyperlipidemia, stroke, anaemia, chronic obstructive pulmonary disease, pulmonary hypertension, preoperative atrial fibrillation, peripheral artery disease), preoperative ACEI, ARB, beta-blockers, loop diuretics, aspirin, and spironolactone use.
Other: surgery-related parameters — 1. surgery type, surgery duration, CPB duration, aortic cross-clamp duration, blood loss, intraoperative fluid infusion, intraoperative urine output, intraoperative blood transfusion, intraoperative anesthetics and vasoactive medications.
  2. duration of mechanical ventilation, duration of vasopressor support, postoperative acute kidney injury incidence and CRRT initiation, major bleeding, deep sternal wound infection/mediastinitis, surgical re-intervention, ICU LOS, hospital LOS, postoperative stroke, complications up to 30 days after surgery, 30-day inpatient mortality, survival status at discharge, and one year follow-up.
  3. a composite endpoint of major complications after surgery defined as at least one of the following: death, prolonged ventilation (>24 h), stroke, severe AKI, deep sternal wound infection, and reoperation for any reason.
Other: POD assessments — Assessments of POD during the first 7 days postoperatively.
Other: collection of biological (laboratory) parameters — 1. WBC, CRP, IL-6, IL-10, IL-1β, TNF-α, serum Amyloid A, procalcitonin, catecholamines, cortisol, SOD, HIF-1α;
  2. BDNF, S-100β protein, NSE;
  3. CK-MB, NT pro-BNP, BNP, high-sensitivity troponin level;
  4. hemoglobin, hematocrit, sodium, arterial lactate, and liver enzymes.
Other: collection of hemodynamic parameters — 1. blood pressure, heart rate, CVP;
  2. CO, CI, SV, SVI,SVV;
  3. intra-abdominal pressure;
  4. vasoactive drug doses in the first hour in the ICU.
Other: collection of echocardiographic parameters and venous ultrasound assessments — (1) Left ventricle systolic function, including LVOT, LVEF, MPI; left ventricular diastolic function, including mitral flow-derived Doppler indices, pulmonary vein Doppler indices. (2) Right ventricular systolic function, including TAPSE. Right ventricular diastolic dysfunction, inferred from an abnormal hepatic vein flow (systolic velocity < diastolic velocity) in the absence of a dysrhythmia or pacing. (3) Inferior vena cava (IVC) measurements. (4) Hepatic vein Doppler parameters. (5) Portal vein Doppler parameters. (6) Renal vein Doppler parameters.
Other: collection of parameters monitoring on the central nervous system — 1. Regional cerebral oximetry.
  2. Brain wave patterns.
  3. Optic nerve sheath diameter.

SUMMARY:
Postoperative delirium (POD) is an acute brain dysfunction characterized by inattention, impaired consciousness, and cognitive and orientation disturbances, and is a common complication after cardiac surgery. The high incidence of up to 52% of POD in cardiac surgery patients lead to a range of adverse clinical outcomes.The brain tissue is enclosed in a rigid anatomical structure; when there is an obstruction to venous return from the brain, intracranial pressure can increase, and blood supply to the brain tissue can decrease, leading to central nervous system dysfunction.

Systemic venous congestion can occur when there is right heart dysfunction or excessive volume load. When right heart failure and/or volume overload occurs, changes in right atrial pressure are transmitted to the venous system of organs throughout the body, with dilatation of the inferior vena cava (IVC), obstruction of blood return from the hepatic, portal, and renal veins, and abnormal venous flow signals and altered ultrasound Doppler flow patterns.

The primary objective of this prospective cohort study is to explore if intraoperative systemic venous congestion is associated with POD after cardiac surgery. This study will also investigate the relationship between intraoperative systemic venous congestion and postoperative complications, and the relationship between each separate venous congestion and POD after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled to undergo elective cardiac surgery via a midline thoracic incision;
2. ≥18 years;
3. A preoperative MMSE score>23, without consciousness or language barriers, capable of cooperating with neurological examinations, cognitive function tests, and other assessments of neurological function.

Exclusion Criteria:

1. Contraindications for TEE;
2. Emergency cardiac surgery;
3. Major vascular surgery;
4. Redo cardiac surgery;
5. Severe infection requiring continuous antibiotic therapy;
6. Severe preoperative heart failure with left ventricular ejection fraction < 30%;
7. A critical preoperative state (mechanical circulatory support, extracorporeal membrane oxygenation, current renal replacement therapy, mechanical ventilation, or cardiac arrest necessitating resuscitation);
8. Multi-organ dysfunction;
9. Known conditions that may interfere with the assessment or interpretation of hepatic vein, portal vein blood flow (such as liver cirrhosis or portal vein thrombosis) or the renal vein blood flow (such as urinary tract obstruction);
10. Planned cardiac transplantation or ventricular assist device implantation;
11. Pregnancy;
12. Insufficient ultrasonographic imaging;
13. Restarting CPB after first CPB cessation during surgery;
14. Requirement for cardiac assist devices (ECMO, IABP, or ventricular assist device) after CPB intraoperatively;
15. Neurological or psychiatric diagnoses that may affect cognitive performance or cognitive testing;
16. Documented delirium before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo elective cardiac surgery
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium after surgery | 7 days after surgery
  Postoperative delirium (POD) is assessed daily using Confusion Assessment Method for Intensive Care Unit (CAM-ICU) or CAM. POD is assessed by formally trained anesthesiologists twice daily from postoperative day 1 to day 7, with assessments conducted in the morning (08:00-10:00) and the afternoon (18:00-20:00). If a positive result is obtained at any time within the first 7 postoperative days, assessments will stop and the case will be recorded as POD.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Zhang, MD, Principal Investigator — The Department of Anesthesiology, The Affiliated Hospital of Yangzhou University, Yangzhou University
Locations (1):
- No. 368 Hanjiang Middle Road, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No